CLINICAL TRIAL: NCT03624842
Title: Expanded Access With Trappsol(R) Cyclo(TM) for an Individual Patient With Late Onset Alzheimer's Disease
Brief Title: Expanded Access With Trappsol(R) Cyclo (TM) for an Individual Patient With Late Onset Alzheimer's Disease
Status: No longer available | Type: Expanded Access
Sponsor: Cyclo Therapeutics, Inc. (Industry)
Collaborators: Kerwin Research Center, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: CTDH-AD-EA-001
Record Dates: First submitted 2018-08-06; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Late Onset Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Trappsol (R) Cyclo (TM)

SUMMARY:
To afford urgent access to a potential-disease modifying treatment, Dr. Diana Kerwin, in partnership with CTD Holdings, the manufacturer of Trappsol (R) Cyclo(TM), will administer the product to a patient with Alzheimer's Disease who has no other disease-modifying treatment options.

DETAILED DESCRIPTION:
Trappsol(R) Cyclo(TM) will be administered via intravenous (IV) infusion. The initial dose will be 500 mg/kg (T=Day 0). Subsequent dosing is anticipated to increase over 9 months, with all subsequent doses given monthly at the maximum dose determined by tolerability, lack of toxicity or adverse event, pharmacokinetic analysis and patient preference. So long as the overall risk/benefit profile favors continued dosing, the patient will continue to receive Trappsol (R) Cyclo (TM) for a minimum of 12 months, if not perpetually.

Risk/benefit assessments will include:

* Vital signs, ECG and laboratory parameters (CBC, chemistry panel, hematology, urinalysis, lipids, coagulation)
* Brain MRI without gadolinium for safety monitoring
* Amyloid and Tau PET (positron emission tomorgraphy) imaging
* Adverse Events
* Mini-mental status score
* Digital Cognition Technologies (DCT) Clock
* Changes in blood biomarkers
* Pharmacokinetic data

ELIGIBILITY:
Inclusion Criteria: Patient with Alzheimer's Disease who continued to decline neurologically and had no other treatment options with intent to halt progression available. All other medical conditions stable & well-managed.

-

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Diana R Kerwin, MD, Principal Investigator — Kerwin Research Center